CLINICAL TRIAL: NCT05013047
Title: Impact of the Covid19 Pandemic on the Organization of Healthcare in France
Brief Title: Impact of the COVID-19 Pandemic on the Organization of Healthcare in France
Acronym: IRIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-13
Record Dates: First submitted 2021-08-18; First posted 2021-08-19 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The 2020 COVID-19 pandemic, which began spreading on January 24, 2020 in France, has required a profound and rapid reorganization of the health system, based in particular on internal hospital reorganizations of front-line establishments, deprogramming of non-urgent activities, and transfers of non-covid19 patients to 2nd line facilities. Beyond the immediate impact on the management of patients infected with COVID-19, this reorganization may have reduced the capacity of management for patients requiring urgent or semi-urgent intervention, or may have postponed some necessary care. The isolation of patients at home may also have resulted in lower compliance to therapy and medical treatments and may have contributed to decompensation.

At the end of this crisis, the different organizational responses in France should be evaluated to identify the consequences and the areas for improvement in order to be prepared for future exceptional health situations. This investigation on healthcare systems confronted to an exceptional health situation thus seeks to determine if the profound reorganizations implemented during this health crisis have indirect effects on the performance of care, in particular if there is a destabilization of the care systems (emergency, semi-emergency and chronic), a loss of chance for the patients and if innovative care paths have emerged.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one of these three types of chronic diseases (Prevention Quality Indicators of the Agency for Healthcare Research and Quality): heart failure, diabetes, chronic obstructive pulmonary disease.
* All French adult patients suffering from the studied chronic diseases, covered by the Health Insurance and living in metropolitan France are included.

Exclusion Criteria:

* Patients under 18 years of age or with incomplete or inconsistent data on the "Système National des Données de Santé", or with a symptomatic COVID-19 diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients without a symptomatic COVID-19 diagnosis, monitored for chronic disease in the French health care system.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess the effect of pandemic COVID-19 on medication compliance in patients with chronic disease | Measured by trimesters (from March 2019 to February 2021)
  Combined chronic drug coverage rate calculated on a three-monthly basis (average of the coverage rates for each drug)

SECONDARY OUTCOMES:
Evaluate the effects of pandemic and lock-down on the risk of decompensation in patients with chronic disease. | 6 months period
  Occurrence of at least one hospitalization for acute decompensation during each of the 6-month periods studied (exposed or not to pandemic and lock-down).

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France